CLINICAL TRIAL: NCT02462330
Title: Effect of Intramyocardial Mesenchymal Stem Cells Injection in Patients With Chronic Ischemic Cardiomyopathy and Left Ventricular Dysfunction Guide by NogaStar XP System Catheter.
Brief Title: Administration of Mesenchymal Stem Cells in Patients With Chronic Ischemic Cardiomyopathy (MESAMI2)
Acronym: MESAMI2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10 142 01
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Chronic Myocardial Ischemia
Keywords: Mesenchymal stem cells; ischemic cardiomyopathy; NogaStar XP system catheter
MeSH Terms: interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo comparator (Placebo Comparator): injection of human albumin 4%
  Interventions: Drug: Placebo comparator
- Autologous MSC from bone marrow (Experimental): intramyocardial injection of 6.10e7 stem cells
  Interventions: Drug: Autologous MSC from bone marrow

INTERVENTIONS:
Drug: Autologous MSC from bone marrow — After bone-marrow aspiration by an authorized person, MSCs were isolated and cultured during 17±2 days by the French Blood Establishment. Then, patients receive intramyocardial injections of MSCs using the electromechanical NOGA-XP system.
  Other Names: mesenchymal stem cells
  Arms: Autologous MSC from bone marrow
Drug: Placebo comparator — injections of human albumin
  Other Names: Human Albumin
  Arms: Placebo comparator

SUMMARY:
Stem cell therapy is an emerging treatment for cardiovascular disease but the best cell type and delivery method remain to be determined. Pre-clinical studies demonstrated improvement of cardiac function by Mesenchymal stem cells (MSC) therapy in particular by their paracrine and immunosuppressive properties. Investigators initiated the MESAMI program by the bicentric pilot phase and highlighted the safety and feasibility of intramyocardial injections of MSCs from bone marrow in patients with chronic ischemic cardiomyopathy and left ventricular dysfunction, guide by the NOGA-XP system. The MESAMI program continues with the phase 2, multicenter, double-blind, randomized, placebo-controlled trial.The aim of this phase 2 study is to demonstrate a functional improvement, measuring peak VO2, at 3 months between the cell therapy group and the placebo group.

DETAILED DESCRIPTION:
Ischemic cardiomyopathies are a leading cause of death in both men and women. During the last decade, treatments for heart failure have evolved, but their purpose is to improve symptoms and prevent aggravation of the disease. Current research is focusing on the development of cell-based therapies using different sources of stem cells which can provide trophic and paracrine support or even replace dying cells with new ones. A specific form of stem cells, called adult mesenchymal stem cells (MSCs), has shown promise for heart repair. These cells are known for their ability to secrete paracrine factors and their immunosuppressive properties. The MESAMI 2 study will evaluate the efficacy of MSCs injection directly into the heart to repair and restore heart function in people with chronic ischemic heart failure using NOGA-XP system.

This phase 2 study is a prospective, multicenter, double-blind, randomized, placebo-controlled trial. A total of 90 patients will be randomized in 2 arms to receive intramyocardial injection of MSCs or placebo. Patients will be followed up for 13 months. Bone marrow will be collected and immediately transported to the French Blood Establishment for MSC isolation and expansion. Patients will receive intramyocardial injection of MSCs or placebo during a left heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Patient who signed the informed consent,
* Chronic stable ischemic cardiomyopathy for at least one month with a NYHA Class II-IV and/or -Angina pectoris CCS Class III or IV,
* Not a candidate for revascularization by coronary artery by-pass surgery or angioplasty,
* Left ventricular function ≤45%,
* Presence of ischemia or myocardial viability on the myocardial perfusion imaging,
* VO2 max≤ 20 ml/min/kg,
* Optimal medical therapy,
* Optimal interventional therapy (Implantable Cardiovertor Defibrillator, effort rehabilitation).

Exclusion criteria:

* Pregnancy or breastfeeding,
* Acute coronary syndrome or myocardial infarction during the last 3 months,
* Revascularization (PCI or CABG), or cardiac resynchronization during the last 3 months,
* Further revascularization planned for the next 30 days,
* LVEF >45%,
* Left intraventricular Thrombus and / or ventricular aneurysm detected by transthoracic echocardiography,
* Wall thickness in the target region <8 mm as determined by echocardiography,
* Critical Limb Ischemia stages 3 or 4,
* Inability to achieve a VO2 test,
* Not feasible peripheral arterial access for percutaneous procedure,
* Aortic stenosis (<1cm²) or aortic insufficiency (> 2 +),
* Patients with transplanted organ,
* Chronic renal failure with creatinemia ≥ 250 µmol/L,
* Severe hepatic dysfunction,
* Chronic atrial fibrillation,
* Decompensated heart failure,
* Uncontrolled Ventricular arrhythmias,
* Indication of cardiac resynchronization by multisite pacemaker or cardiac resynchronization during the last 3 months,
* Obesity preventing bone marrow aspiration or manual compression of the puncture area after bone marrow collection,
* Active uncontrolled infection
* Immuno-modulator treatment (ciclosporin, mycophenolate, mycophenolate mofetil, azathioprine, tacrolimus, anthracyclines, neupogen, hydrea, etanercept interferons, prednisolone, methylprednisolone, colchicine),
* History of cancer in the last 5 years,
* Hemopathy, hematopoietic disease,
* Haemorrhagic syndrome,
* Chronic or progressive disease that may alter the prognosis within 3 months,
* Positive serologies for Human immunodeficiency virus (HIV1-2), HTLV-1 (human T-cell lymphotrophic virus) and 2, HBV (hepatitis B virus) or HCV (hepatitis B virus).
* Allergic to xylocain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Change in VO2max | 3 months
  Change in VO2max (or peak VO2) before injection and at 3 months post injection.

SECONDARY OUTCOMES:
Left ventricular viability | Before injection and at 3, 6 and 12 months
  MRI
NYHA/CCS class | Before injection and at 3, 6 and 12 months
  Change on class
Quality of life (Minnesota questionnaire) | Before injection and at 3, 6 and 12 months
  Change on quality of life test score
VO2 max | At 6 and 12 months
  Change in VO2max (or peak VO2) at 6 and 12 months post injection.
6'walking-test | Between 3 and 12 months
  Distance to walk test
Echocardiography | Before injection and at 3, 6 and 12 months
  Volume of myocardium and measurement of ejection fraction
Myocardial perfusion imaging | Before injection and at 3, 6 and 12 months
  Efficacy of the cell therapy on LVEF
BNP blood test | Before injection and at 3, 6 and 12 months
  Change of the BNP blood test at 3, 6 and 12 months

OTHER OUTCOMES:
Adverse event related to cell administration | 12 months
Complication related to cell administration | 12 months
Control of the implantable cardioverter defibrillator | 12 months
Analysis of major cardiovascular events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerôme Roncalli, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (6):
- France (6):
  - University hospital of Henri Mondor, Créteil
  - University hospital of Grenoble, Grenoble
  - University hospital of Lille, Lille
  - University hospital of Nantes, Nantes
  - University hospital of Pitié-Salpêtrière, Paris
  - Cardiology Department of Rangueil Hospital - Rangueil Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No